CLINICAL TRIAL: NCT05150899
Title: Comparative Study Between Use of Alpha Blocker Versus Alpha Blocker and Antihistaminic in Management of Acute Renal Colic Prevent Pain Recurrence and Increase Expulsion Rate of Ureteric Stone ≤ 1cm
Brief Title: Role of Antihistaminic in Acute Renal Colic Prevent Pain Recurrence and Expulsion of Ureteric Stone ≤ 1cm
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Kamel Abdel Rahman, Director, Assiut University
Other Study IDs: antihistaminic in renal colic
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Renal Colic; Ureter Stone
MeSH Terms: conditions — Renal Colic; Ureterolithiasis | interventions — Tamsulosin; Capsules; fexofenadine; Tablets

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Tamsulosin 0.4mg: group A receive Tamsulosin 0.4mg in combination of NSAI drug if patient present with colic, if not in renal colic at bed time Tamsulosin 0.4mg with analgesic on demand.
  Interventions: Drug: Tamsulosin Hcl 0.4Mg Cap
- fexofenadine 180 mg in combination of Tamsulosin 0.4mg: group B receive pheniramine maleate 50mg injection every 12hr for 24 hr in combination of Tamsulosin 0.4mg and NSAI drug then fexofenadine 180 mg in combination of Tamsulosin 0.4mg and NSAI drug on demand if patient present with colic. if not in renal colic at bed time fexofenadine 180 mg in combination of Tamsulosin with NSAI on demand.
  Interventions: Drug: Tamsulosin Hcl 0.4Mg Cap; Drug: fexofenadine 180 mg Oral tablet

INTERVENTIONS:
Drug: Tamsulosin Hcl 0.4Mg Cap — alpha blocker
  Other Names: tamsule
Drug: fexofenadine 180 mg Oral tablet — antihistaminic
  Other Names: telefast
  Groups: fexofenadine 180 mg in combination of Tamsulosin 0.4mg

SUMMARY:
Urolithiasis is one of the most common urological diseases. The risk of stone disease ranges between 5% and 12% worldwide. Ureteric stones account for ≈20% of all urinary tract stones and >70% of the ureteric stones are located in the lower third of the ureter, i.e., distal ureteric stones (DUS). The colicky-type pain in the ureter, an increase in proximal peristalsis through activation of intrinsic ureteral pacemakers may contribute to the perception of pain. Muscle spasm increased proximal peristalsis, local inflammation, irritation, and oedema at the site of obstruction may contribute to the development of pain through chemoreceptor activation and stretching of submucosal free nerve endings. α-adrenergic blockers, anti-inflammatory drugs, antihistaminic and calcium channel blockers, which have a relaxant effect on the ureteric smooth musculature. The presence of histamine receptors in the ureter have been presented in various studies. The histamine-1 (H1) receptors have been shown to have a wide distribution Histamine, which is secreted from the mast cells, causes strong peristaltic contractions in the ureter. alpha adrenoreceptor antagonists (i.e., tamsulosin) have been employed in the treatment of ureteric colic due to smooth muscle relaxation so their potential ability to increase stone passage, reduce pain medication use and reduce urologic interventions. According to the currently accepted view, renal colic management starts with NSAI drugs also NSAI has role in decrease inflammation and oedema and increase expulsion rate . in this study we will compare the use of alpha blocker versus alpha blocker and antihistaminic in management of acute renal colic prevent pain recurrence and increase expulsion rate of ureteric stone ≤ 1cm, with analgesic use in case of acute stage.

DETAILED DESCRIPTION:
All the patients will be included within inclusion criteria After providing written informed consent, these patients were randomly divided into 2 groups by use of a computer-generated random number table.

1. history taken about patient pain onset, duration and type with scoring the pain by World Health Organization numerical pain score of 0-10.
2. Ultrasonography done to determine if kidney obstructed and grade of obstruction at the day 1 day 15 and day 30.
3. group A receive Tamsulosin 0.4mg in combination of NSAI drug if patient present with colic, if not in renal colic at bed time Tamsulosin 0.4mg with analgesic on demand, group B receive pheniramine maleate 50mg injection every 12hr for 24 hr in combination of Tamsulosin 0.4mg and NSAI drug then fexofenadine 180 mg in combination of Tamsulosin 0.4mg and NSAI drug on demand if patient present with colic. if not in renal colic at bed time fexofenadine 180 mg in combination of Tamsulosin with NSAI on demand.
4. In case of patient presented by acute renal colic the time of administration of treatment recorded and the time of relief pain recorded.
5. CT scan done to ensure urolithiases if no CT done at the first day and after 30 days.
6. Full labs done especially serum creatinine and serum uric acid.

ELIGIBILITY:
Inclusion Criteria:

* Age from 14 to 70 years old.
* Patient with ureteric stone 5-10 MM.
* Patient with acute renal colic presented to emergency with obstructed kidney with urgent MSCT show stone ureter 5-10 MM and patient come without colic with CT showing lower third stone of the same measurement.

Exclusion Criteria:

* Age less than 14 or more than 70.
* Chronically diseased patient cardiac that contraindicated to take PD5I or tamsulosin.
* Only functioning kidney.
* CKD Patient.
* Bilateral ureteric stone.
* urinary tract infection.
* severe refractory pain.
* severe hydronephrosis.
* multiple ureteric stones.
* ischemic heart disease, congestive cardiac failure, or complicated hypertension.
* pregnant or lactating mothers.
* patient refuse medical treatment.
* congenital anomalies.
* previous ureteric surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All cases that fulfil the selection criteria that will be followed up in the department of Assiut university hospital (non-probability sample size) with Confidence Level 90 %, Population Size 10000, Margin of Error 8 % with expected size of 100 patients enrolled in the study. these patients were randomly divided into 2 groups 50 in each group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-11-25 (Estimated); Study Completion 2022-11-25 (Estimated)

PRIMARY OUTCOMES:
Success rate of each treatment in case of patient presented with acute renal colic | 3 weeks
  (% of patients show relief of the pain).
Duration of relieve of the symptoms | in 24 hours
  relieve of renal colic
Rate of recurrence of pain and if need analgesic | 3 weeks
  how many times pain come again
Numbers of patients showing expulsion of stone | 3 weeks
  how many people stone expulsed during treatment
Number of patients underwent URS and duration taken from start of treatment | 3 weeks
  patient with persistent pain
Rate of complication from treatment | 3 weeks
  any side effect from treatment
Rate of hospital admission and number of admissions. | 3 weeks
  due to persistent pain
Rate of drop out from the study due to complication or noncompliance. | 3 weeks
  patient exit from study

CONTACTS AND LOCATIONS:
Overall Officials: adel kurkar, MD, Principal Investigator — Assiut University; mostafa kamel, demonstrator, Principal Investigator — Assiut University; ahmed eltaher, MD, Study Chair — Assiut University; ahmed elbadry, MD, Study Chair — Assiut University; ahmed abdelhameed, MD, Study Chair — Assiut University; rabee gadelkareem, MD, Study Chair — Assiut University; hosney behnsawy, MD, Study Chair — Assiut University; mohamed zarzour, MD, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bader MJ, Eisner B, Porpiglia F, Preminger GM, Tiselius HG. Contemporary management of ureteral stones. Eur Urol. 2012 Apr;61(4):764-72. doi: 10.1016/j.eururo.2012.01.009. Epub 2012 Jan 14. PMID 22266271
- [Result] Coll DM, Varanelli MJ, Smith RC. Relationship of spontaneous passage of ureteral calculi to stone size and location as revealed by unenhanced helical CT. AJR Am J Roentgenol. 2002 Jan;178(1):101-3. doi: 10.2214/ajr.178.1.1780101. PMID 11756098
- [Result] Hollingsworth JM, Rogers MA, Kaufman SR, Bradford TJ, Saint S, Wei JT, Hollenbeck BK. Medical therapy to facilitate urinary stone passage: a meta-analysis. Lancet. 2006 Sep 30;368(9542):1171-9. doi: 10.1016/S0140-6736(06)69474-9. PMID 17011944
- [Result] Giuliano F, Uckert S, Maggi M, Birder L, Kissel J, Viktrup L. The mechanism of action of phosphodiesterase type 5 inhibitors in the treatment of lower urinary tract symptoms related to benign prostatic hyperplasia. Eur Urol. 2013 Mar;63(3):506-16. doi: 10.1016/j.eururo.2012.09.006. Epub 2012 Sep 11. PMID 23018163
- [Result] Gratzke C, Uckert S, Kedia G, Reich O, Schlenker B, Seitz M, Becker AJ, Stief CG. In vitro effects of PDE5 inhibitors sildenafil, vardenafil and tadalafil on isolated human ureteral smooth muscle: a basic research approach. Urol Res. 2007 Feb;35(1):49-54. doi: 10.1007/s00240-006-0073-1. Epub 2006 Nov 11. PMID 17102958
- [Result] Kumar S, Jayant K, Agrawal MM, Singh SK, Agrawal S, Parmar KM. Role of tamsulosin, tadalafil, and silodosin as the medical expulsive therapy in lower ureteric stone: a randomized trial (a pilot study). Urology. 2015 Jan;85(1):59-63. doi: 10.1016/j.urology.2014.09.022. PMID 25530364
- [Result] Ugaily-Thulesius L, Thulesius O. The effects of urine on mast cells and smooth muscle of the human ureter. Urol Res. 1988;16(6):441-7. doi: 10.1007/BF00280026. PMID 2466358
- [Result] Hollingsworth JM, Canales BK, Rogers MA, Sukumar S, Yan P, Kuntz GM, Dahm P. Alpha blockers for treatment of ureteric stones: systematic review and meta-analysis. BMJ. 2016 Dec 1;355:i6112. doi: 10.1136/bmj.i6112. PMID 27908918
- [Result] Shokeir AA. Renal colic: new concepts related to pathophysiology, diagnosis and treatment. Curr Opin Urol. 2002 Jul;12(4):263-9. doi: 10.1097/00042307-200207000-00001. PMID 12072644